CLINICAL TRIAL: NCT00294242
Title: Does Routine Membrane Sweeping in Uncomplicated Term Pregnancies Increase the Rate of Prelabour Rupture of Membranes
Brief Title: Safety Study of Membrane Sweeping in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6H06
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy; Prelabor Rupture of Membranes
Keywords: pregnancy; membranes sweeping; prelabor rupture of membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

ARMS (2):
- Membrane Sweep (Active Comparator): Weekly membrane sweeping performed for the duration of the pregnancy after 38 0/7 weeks gestational age
  Interventions: Procedure: Membrane Sweep
- No Membrane Sweep (Experimental): No membrane sweeping conducted for the duration of the pregnancy after 38 0/7 weeks gestational age
  Interventions: Procedure: No Membrane Sweep

INTERVENTIONS:
Procedure: Membrane Sweep — Weekly Membrane Sweep
  Arms: Membrane Sweep
Procedure: No Membrane Sweep — No Membrane Sweep
  Arms: No Membrane Sweep

SUMMARY:
The purpose of this study is to determine if routine membrane sweeping in uncomplicated term pregnancies increases the rate of pre-labor rupture of membranes.

DETAILED DESCRIPTION:
The question of routine membrane sweeping and prelabor rupture of membranes has not been specifically addressed in a randomized control trial. A meta analysis of membrane sweeping found ten publications which analyzed this question as a secondary outcome, though none of these studies sought to analyze PROM in their objectives. This meta analysis found the relative risk of prelabor rupture of membranes to be 1.14 with membrane sweeping, however the confidence interval was 0.89 to 1.45 making the finding not significant. Despite this, we feel that a study to specifically address this issue is warranted. The largest study in the meta analysis (and the only one with a statistically significant difference on its own) did find a significant risk of PROM. The studies in the meta analysis vary greatly in their incidence of PROM, ranging from 2-39% in the membranes sweeping group and 2-26% in the control groups. This wide variation, the fact these studies were not primarily designed to compare PROM rates, and the reported 8-10% PROM in other texts and studies gives question to the ability of this meta analysis to detect a difference in PROM rates between the two groups. As the effect of membrane sweeping on PROM may influence clinicians attitudes toward this intervention, further specific research is warranted.

Our Objective are:

1. To determine the rate of prelabor rupture of membranes in uncomplicated term pregnancies undergoing routine membrane sweeping versus those without intervention. For the purpose of this study, PROM is defined as the confirmation of ruptured amniotic fluid with uterine contractions less than 10 minutes apart.
2. To determine the impact of membrane sweeping on successful labor induction for post datism and pregnancies going past 41 weeks
3. To determine the impact of membrane sweeping and PROM with clinical variables

Patients will be randomized by a computer generated randomizer to either receive membrane sweeping or vaginal exam without membrane sweeping. Patients will receive either membrane sweeping or vaginal exam without membrane sweeping at each weekly visit from 38 weeks gestation onwards. Patients in the no intervention group will receive no cervical evaluation unless clinically indicated. Patients in the membrane sweeping group will have a finger placed into the cervical os, the finger will be rotated in a 360 degree fashion which will separate the amniotic membranes from by a circular motion. Patients in this group whose cervix is not open enough to have the membranes swept will have it gently stretched and if the cervix is closed it will be gently massaged to stimulate the release of prostaglandins (1). Due to the nature of the intervention, it is not possible to blind the physician who is performing the vaginal exam to which group the patient is in. However, the admitting and delivering physicians will be blinded to the group allocations. This will minimize bias. Such blinding will be done by having a patient identifier code in the chart which the clinic physicians will use to access the randomizer online for determination of which exam to perform. Admitting and delivering physicians will not access this code. Between 38 and 42 weeks gestation, clinical data from each prenatal visit will be kept to include patient age, gestational age, parity, race, cervical exam, post-graduate year level of physician or if the provider is a midwife or attending staff, and whether or not membrane sweeping was performed. In Labor and Delivery data will then be collected on gestational age at delivery, indication for admission, inductions, reason for induction, estimated gestational age at delivery, PROM, cervical exam at admission, Bishop's score on admission, labor outcomes, route or delivery, pregnancy complications, neonatal complications, GBS status, and NICU admissions. PROM as an indication for admission will be confirmed by nitrazine testing, ferning test, and speculum examination. Two of the three tests must indicate PROM for the patient to be given the diagnoses of PROM. PROM will be defined as the above positive testing with contractions more than 10 minutes apart at the time of rupture of membranes. If the PROM occurred just prior to the examination, this assessment will be made on the tocometer. If the PROM occurred prior to the patient presenting to Labor and Delivery, this assessment will be based on the patient's subjective assessment of her contractions at the time of membrane rupture. Labor is defined as regular contractions leading to cervical change. The frequency of contractions required to cause cervical change varies from patient to patient, however for the purpose of this study the patient will be considered to have SROM (spontaneous rupture of membranes due to labor) if contractions are more frequent than every 10 minutes. Patients will be analyzed on an intent to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated, singleton pregnancies
* candidates for vaginal delivery
* 38 to 42 weeks estimated gestational age

Exclusion Criteria:

* multiple gestation
* placenta previa
* placental abruption
* pre-gestational or gestational diabetes
* chronic or gestational hypertension
* pre-eclampsia
* pregnancy before 38 weeks gestation
* any pregnancy with an indication for induction other than impending post dates
* any pregnancy not planning of vaginal delivery
* history or preterm labor or prelabor rupture of membranes
* vasa previa
* cervical dilation 3cm or greater upon entry to study
* active cervical infection
* third trimester vaginal bleeding
* significant maternal mullerian anomalies
* severe fetal anomalies
* active genital herpes infection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Prelabor membranes rupture | 3 weeks
  Rates of prelabor rupture of membranes

CONTACTS AND LOCATIONS:
Overall Officials: Micah J Hill, D.O., Principal Investigator — United States Army
Locations (1):
- Tripler Army Medical Center, Tripler AMC, Hawaii, United States

REFERENCES:
- [Background] 1. Bulware et al. Membrane sweeping for induction of labor. The Cochrane Database for induction of labor 2005, 2 (no page number) 2. Magann et al. Can we decrease postadtism in women with an unfavorable cervix and a negative fetal fibronectin test result at term by serial membrane sweeping? Am J Obstet Gynecol 1998, 179(4): 890-894 3. CammuH, Haitsma V. Sweeping membranes at 39 weeks in nulliparous women: a randomized controlled trial. Brit J Obstet Gynecol 1998: 105(1): 41-4 4. Boulvain et al. Does sweeping of the membranes reduce the need for formal induction of labour? A randomized controlled trial. Brit J Obstet Gynecol. 1998, 105(1): 34040 5. Allott HA, Palmer CR. Sweeping the membranes: a valid procedure in stimulating the onset of labour? Brit J Obstet Gynecol 1993, 100(10): 889-90 6. Wong et al. Does sweeping of membranes beyond 40 weeks reduce the need for formal incution of labour? Brit J Obstet Gynecol 2002, 109(6): 632-6 7. Sweeping of the membranes is an effective method of induction of labor in prolonged pregnancy: a report of a randomized trial. Brit J Obstet Gynecol 1992, 100(10): 898-903 8. McColgin et al. Partuitional factors associated with membrane stripping. Am J Obstet Gynecol. 1993, 169(1): 71-77 9. Keirse et al. Chronic stimulation of uterine prostaglandin synthesis during cervical ripening before the onset of labor. Prostaglandins, 1983, 25(5): 671-82 10. Goldenberg et al. Stretching of the cervix and stripping of the membranes at term: a randomized controlled study. Eur J Obstet Gynecol 1996, 66(2): 129-32 11. Tannirandorn Y, Jumrustanasan T. A comparative study of membrane stripping and nonstripping for induction of labor in term pregnancy. J Med Assoc of Thailand 1999, 82(3): 229-32 12. Williams Obstetrics. McGraww-Hill Companies. New York, NY. 2000, 440-1. 13. Maternal-Fetal Medicine. WB Saunders. Philedelphia, PA. 1999. 644-5. 14. Induction of Labor. Compendium of Selected Publications. ACOG Practice Bulletin. Nunmber 10, Nov 1999, 437-482. Merck, Washington, DC 2005. 15. De Grace et al. Induction of labour with a favourable cervix and/or pre-labour rupture of membranes. Clin Obstet Gynaecol. 2003 Oct;17(5):795-809. 16. Misoprostol versus expectant management in premature rupture of membranes at term. Brit Jour Obstet Gynecol. 2005 Sep;112(9):1284-90. 17. Permature Rupture of Membranes. ACOG Practice Bulletin. Number 1, June 1998, pgs 697-705. 18. Sahraoui W. et al. Management of pregnancies beyond forty-one week's gestation with an unfavorable cervix. J Gynecol Obstet Biol Reprod (Paris). 2005 Sep;34(5):454-62.
- [Derived] Hill MJ, McWilliams GD, Garcia-Sur D, Chen B, Munroe M, Hoeldtke NJ. The effect of membrane sweeping on prelabor rupture of membranes: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1313-9. doi: 10.1097/AOG.0b013e31816fdcf3. PMID 18515514